CLINICAL TRIAL: NCT03034486
Title: A Single Sequence, 3-period, Multiple-dose Study to Evaluate the Pharmacokinetics of D565 and the Drug Effect of D565 on Pharmacokinetic Characteristics of D930 in Healthy Male Volunteers
Brief Title: The Pharmacokinetics of D565 and the Drug Effect of D565 on Pharmacokinetic Characteristics of D930
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171DDI16019
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single sequence, 3-period (Experimental)
  Interventions: Drug: D930, D565

INTERVENTIONS:
Drug: D930, D565 — Period 1: D565 administered 1 time for one day/ Period 2: D930 administered 3 time per day for 9 days/ Period 3: D565(1 time per day) with D930(3 time per day) administered for 9days

SUMMARY:
This study is a single sequence, 3-period, multiple-dose study to evaluate the pharmacokinetics of D565 and the drug effect of D565 on pharmacokinetic characteristics of D930 in healthy male volunteers.

DETAILED DESCRIPTION:
This study is a single sequence, 3-period, multiple-dose study to evaluate the pharmacokinetics of D565 and the drug effect of D565 on pharmacokinetic characteristics of D930 in healthy male volunteers.

Subjects will receive D565 just one time on period 1 for evaluate the pharmacokinetics. And afterward, subjects will receive multiple dose of D930 for 9 days, and D565 with D930 for 9 days to evaluate the drug effect on period 2 and 3.

When period 1 finished, there are 3 days of washout period, but between period 2 and 3, there is no washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male older than 19 years and younger than 55 years at the time of screening
2. BMI 18.0~30.0(kg/m2) and body weight more than 55kg
3. Subject who has no chronic disease within last 3 years, no symptoms or pathological findings
4. Suitable subject who is determined by laboratory tests that hematology test, blood chemistry, urinalysis test according to the characteristics of the drug and 12-lead ECG at the time of screening
5. Subject who fully understand the purpose and content of clinical trials, characteristic of the drug after in-depth explanation, decided to join the clinical trials by their will and signed inform consent
6. Subject who has will and ability to participate in clinical trials

Exclusion Criteria:

1. Subject who has a history of clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, psychiatric, neurological, allergic or ophthalmic diseases (except for asymptomatic seasonal allergies not treated at the time of single administration) or who has a following history

1. Patients with liver failure or severe renal disease(CCr < 30ml/min) and cardiovascular patient (CCr is calculated by Cockroft and Gault formula)
2. Patients with acute occlusion angle glaucoma
3. Patients with a history of kidney stones
4. Patients with a history of chronic corneal injury and ophthalmic surgery
5. Patients with decreased endothelial cell count
6. Patients with renal tubular cells immature or with perchloric acidosis
7. Patients receiving MAO inhibitor
8. Patients taking antidepressants that affect noradrenaline delivery
9. Patients with depression, cerebral impairment or coronary artery disease, Raynode phenomenon, standing hypotension, and obstructive thromboangitis
10. Patients with bronchial asthma or history of asthma

2. Those who meet the following criteria on ophthalmological examination or test

1. A person with a history or suspected symptom of visual organs diseases including keratitis, iritis, uveitis, retinitis, dry eye syndrome, and strabismus.
2. Those who have had previous ophthalmic surgery or have undergone ophthalmic laser surgery within 6 months
3. Those whose corrected visual acuity measured at screening is 20/40 (acupuncture visual acuity chart 0.5) or less.
4. Those who have experienced side effects after wearing contact lenses, or who have worn contact lenses since the last month, who can not comply with the prohibition of wearing contact lenses during clinical trials
5. Others who have abnormal findings on ophthalmic examination

3. Patients with a history of gastrointestinal disorders (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (excluding simple cecal surgery or hernia surgery) that may affect the absorption of pharmaceuticals for clinical trials

4. Clinical laboratory test results showing the following values

1. ALT or AST> 2 times upper limit of normal range
2. eGFR <60 mL / min / 1.73m2 calculated by the Modification of Diet in Renal Disease (MDRD)

5. When the systolic blood pressure is less than 100 mmHg or more than 150 mmHg or diastolic blood pressure is less than 60 mmHg or not less than 100 mmHg

6. Those who have received medication within 3 months prior to the first administration of the clinical trial drug by participating in other clinical trials or bioequivalence studies (However, the ending date of participation in the examination shall be the last day of medication.)

7. Those who have a history of drug abuse within the first year of screening

8. Persons who have been drinking continuously (21 units / week, 1 unit = 10 g of pure alcohol) within 6 months of the first dose or who can not abstain during the trial Example> Beer 5 ° 1 cup (250 ml) = 10 g, Soju 20 ° 1 cup (50 ml) = 8 g, Wine 12 ° 1 cup (125 ml) = 12 g

9. Those taking medication known to induce or inhibit drug metabolizing enzymes within 30 days prior to the first administration of clinical trial medication

10. A person taking any prescribed medicinal product or herbal medicine within 2 weeks of the first day of administration or taking or applying any OTC drug or vitamin preparation including artificial tears within 1 week (However, depending on the testee's judgment, other conditions may be appropriate to participate in the clinical trial)

11. Those who have received a whole blood donation within 2 months before the first administration of the drug for clinical trial, or have received a blood donation and blood transfusion within 1 month

12. Persons with hypersensitivity or clinically significant hypersensitivity reactions to medicinal products for use in clinical trials or drugs containing the same class of ingredients (eg. latanoprost, benzalkonium chloride)

13. Those who are not willing or able to comply with the lifestyle guidelines described in this Protocol,

14. An average of 10 smokers per day over the past three months or who can not quit smoking 48 hours before the first dose

15. Those who are planning to become pregnant during the trial period or who are not planning to use a reliable contraceptive method (Eg, use of contraceptives and transplants or intrauterine devices, infertility procedures (vasectomy, tubal ligation, etc.), blockage (condoms and spermicide), vaginal septa, vaginal sponges,

16. A person who is found to be unsuitable for clinical trial participation due to other reasons including clinical laboratory test results

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h
Cmax,ss of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h

SECONDARY OUTCOMES:
AUCt of D565 | predose (0 h), 1min, 3min, 5min, 10min, 15min, 20min, 40min, 1, 2, 4 h
Cmax of D565 | predose (0 h), 1min, 3min, 5min, 10min, 15min, 20min, 40min, 1, 2, 4 h
Tmax of D565 | predose (0 h), 1min, 3min, 5min, 10min, 15min, 20min, 40min, 1, 2, 4 h
t1/2 of D565 | predose (0 h), 1min, 3min, 5min, 10min, 15min, 20min, 40min, 1, 2, 4 h
AUCinf of D565 | predose (0 h), 1min, 3min, 5min, 10min, 15min, 20min, 40min, 1, 2, 4 h
Ctrough, ss of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h
Tmax,ss of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h
t1/2 of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h
AUCinf of D930 | predose (0 h), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, Ph.D, Principal Investigator — The Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Seo-gu, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No